CLINICAL TRIAL: NCT01528696
Title: Silver Impregnated Dressings to Reduce Wound Complications in Obese Patients at Cesarean Section
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: University of Michigan (Other)
Collaborators: Cura Surgical (Unknown)
Responsible Party: Principal Investigator, Mark Chames, MD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00037674
Record Dates: First submitted 2012-02-01; First posted 2012-02-08 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Complications; Caesarean Section, Wound
Keywords: Obesity; Cesarean Section; Wound care
MeSH Terms: conditions — Obesity; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Dressing (Placebo Comparator): Obese patients undergoing cesarean section in this arm will receive a standard island-type dressing
  Interventions: Device: Standard Dressing
- Silverlon (Experimental): Obese patients undergoing cesarean section in this arm will receive Silverlon, a silver impregnated dressing
  Interventions: Device: Silverlon

INTERVENTIONS:
Device: Silverlon — Patients will be randomized to either receive a silver dressing. Patients who receive a silver dressing will have that dressing replaced on postoperative day number 2. This will be left in place until the patient is seen for follow up by the visiting nurse.
  All patient will be evaluated by the visiting nurse on postoperative day 4 or 5 and have their wounds photographed. All patients will be contacted for a brief survey 6 weeks postpartum.
  Arms: Silverlon
Device: Standard Dressing — Standard island dressing. Patients who receive a standard dressing will have that dressing removed on postoperative day 2. This will be left in place until the patient is seen for follow up by the visiting nurse.
  Arms: Standard Dressing

SUMMARY:
Obese patients undergoing cesarean section are at high risk for wound complications, which occur in approximately 20% of patients. This is a randomized controlled trial designed to determine whether the risk for wound-related complications can be reduced by covering the incision with a silver-impregnated dressing in the postoperative period.

DETAILED DESCRIPTION:
This study's purpose was to evaluate the effect of a FDA approved silver-impregnated dressing on cesarean wound complications in obese women. It was initiated and 37 women were randomized, but because of logistical barriers, we were unable to gather outcome data either by the intended survey or by chart review. When it became clear that we would be unable to complete the study, recruitment was terminated and further attempts at data gathering were stopped. While a small number of photographs were taken as intended, they were lost due to a technological failure prior to any analysis. Therefore no outcome data could be analyzed. Nonetheless, as patients of the University of Michigan Health System, all research subjects received health care treatment appropriate to their medical condition and circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cesarean section (with or without concurrent tubal ligation)
* Body mass index (based on most recent weight) >=30

Exclusion Criteria:

* Known allergy to silver
* Less than 18 years of age
* Preoperative evidence of current abdominal wall infection
* Contraindication to closure of the skin at time of surgery
* Plan to perform procedures in addition to cesarean section (with or without tubal ligation)
* Patients with previously placed abdominal wall mesh at site of planned surgery
* Inability to participate in medical decision making
* Inability to follow up with the Michigan Visiting Nurses or are unable to return to the University of Michigan Medical Center for staple removal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chames, MD, Principal Investigator — University of Michigan; Angela Liang, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Von Voigtlander Womens' Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Krieger BR, Davis DM, Sanchez JE, Mateka JJ, Nfonsam VN, Frattini JC, Marcet JE. The use of silver nylon in preventing surgical site infections following colon and rectal surgery. Dis Colon Rectum. 2011 Aug;54(8):1014-9. doi: 10.1097/DCR.0b013e31821c495d. PMID 21730792
- [Background] Epstein NE. Do silver-impregnated dressings limit infections after lumbar laminectomy with instrumented fusion? Surg Neurol. 2007 Nov;68(5):483-5; discussion 485. doi: 10.1016/j.surneu.2007.05.045. PMID 17961738
- [Background] Huckfeldt R, Redmond C, Mikkelson D, Finley PJ, Lowe C, Robertson J. A clinical trial to investigate the effect of silver nylon dressings on mediastinitis rates in postoperative cardiac sternotomy incisions. Ostomy Wound Manage. 2008 Oct;54(10):36-41. PMID 18927482
- See also: University of Michigan Department of Obstetrics and Gynecology — http://obgyn.med.umich.edu/
- See also: Cura Surgical — http://ww.curasurgical.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Silverlon: Obese patients undergoing cesarean section in this arm will receive Silverlon, a silver impregnated dressing
  Silverlon: Patients will be randomized to either receive a silver dressing. Patients who receive a silver dressing will have that dressing replaced on postoperative day number 2. This will be left in place until the patient is seen for follow up by the visiting nurse.
  All patient will be evaluated by the visiting nurse on postoperative day 4 or 5 and have their wounds photographed. All patients will be contacted for a brief survey 6 weeks postpartum.
Period: Overall Study
Arm/Group | Standard Dressing | Silverlon
Started | 18 | 19
Hospital Stay (2-5 Days) | 18 | 19
Completed | 0 | 0
Not Completed | 18 | 19
Not completed — See detailed description | 18 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dressing | Silverlon | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience One or More Wound Complications
Description: A composite of cellulitis, wound dehiscence, seroma, hematoma, abscess, and fascial dehiscence from wound evaluation at any point within six weeks, as pulled from the medical record or based on patient report.
Time Frame: 6 weeks
Population: For logistical reasons, we were unable to gather outcome data either by the intended survey or by chart review. When it became clear that we would be unable to complete the study, recruitment was terminated and further attempts at data gathering were stopped. Therefore no outcome data could be analyzed.
Arm/Group | Standard Dressing | Silverlon
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Febrile Morbidity
Description: Febrile morbidity would be measured by number of participants who experienced fever as a sign of infection at 2 days, and overall within 6 weeks of delivery.
Time Frame: 2 days, 6 weeks
Population: as for outcome 1
Arm/Group | Standard Dressing | Silverlon
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Report of Pain Severity and Control
Description: Self Reported pain, on a scale from 1 to 10, where 1 is little pain and 10 is extreme pain
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Standard Dressing | Silverlon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The original intent was to pull adverse event data from the medical record in batches as the study progressed. Because enrollment ceased early with insufficient numbers to draw conclusions, no adverse event data was collected in study. Therefore the 0 numbers affected listed below in serious and other adverse events represent no collected data of adverse events, not a guarantee that no adverse events happened. All participants were under medical care with attending physicians at all times.
Arm/Group | Standard Dressing | Silverlon
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes